CLINICAL TRIAL: NCT04602858
Title: Reactive Balance Training Involving Repeated Trips and Slips in Older Adults: Mechanisms and Long-term Retention
Brief Title: The SafeTrip Study - Step Training to Reduce Falls in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroscience Research Australia (Other)
Collaborators: The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HC190952; U1111-1258-0513 (Other: WHO Universal Trial Number)
Record Dates: First submitted 2020-09-14; First posted 2020-10-26 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Fall; Fall Injury
Keywords: falls; fall prevention; balance; muscle; reflex; reactive balance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reactive Balance Training (Experimental): Participants randomised to the intervention group will initially undertake 3 x 40 min training sessions of reactive balance training over 3 weeks followed by 3-monthly retraining sessions at 3, 6 and 9 months, and final assessment at month 12.
  During the training, participants will be exposed to unpredictable slips and trips whilst they are walking on the Trip and Slip Walkway (Okubo et al. 2019). They will be required to consistently walk at their normal walking pace using our gait regulation protocol (i.e. individually adjusted stepping tiles and metronome). Each training session will involve up to 30 trips and slips which progress in unpredictability.
  Participants will also receive a "Staying active and on your feet" fall prevention booklet containing guidance regarding fall risk factors including exercise, diet, vision, footwear, medications and home safety.
  Interventions: Device: Reactive Balance Training
- Control (Active Comparator): After exposing the control group to one trip and one slip at baseline, participants will then be provided with the "Staying active and on your feet" fall prevention booklet, an educational booklet providing guidance on fall risk factors including exercise, diet, vision, footwear, medications and home safety. The control group will then return for a reassessment after 12 months.
  Interventions: Other: Control

INTERVENTIONS:
Device: Reactive Balance Training — Reactive balance training involves the use of the Trip and Slip walkway that is able to expose participants to unpredictable trips and slips. Trips and slips will occur at random location on the walkway and times within the gait cycle, with the participants receiving 3-monthly retraining sessions along with an educational booklet.
  Arms: Reactive Balance Training
Other: Control — The control intervention will be receiving an educational booklet as part of standard care. The education component will target a variety of fall risk factors and provide strategies to mitigate these risk factors.
  Arms: Control

SUMMARY:
Falls in older people are devastating, widespread, costly and increasing in the aging Australian population. Although falls occur in approximately one third of older adults, certain population groups such as the sarcopenic/frail present with further elevated risk of falls. Many exercise interventions have been trialled but systematic review evidence indicates such programs reduce fall rates by an average of only 20% and encounter issues such as compliance.

Reactive balance training (also called perturbation-based balance training) utilises a task-specific approach to balance training, applying repeated exposure to unpredictable perturbations that mimic balance disturbances experienced in daily life. Evidence suggests 50% reductions in falls might be achievable in a time efficient manner with reactive balance training but more evidence is required.

In this study, ecologically valid, unpredictable trips and slips will be exposed to older people in a safe environment to train their reactive balance. Three 40 min weekly training sessions will be followed by 3-monthly retraining session over one year (40 min x 6 training sessions = 4 hours of training in total). The neuromuscular, physiological, psychological, behavioural effects of the reactive balance training will be comprehensively examined.

ELIGIBILITY:
Inclusion Criteria:

* Older persons - aged 65 years and older
* Community-dwelling
* Ability to walk 500m without rest or use of mobility aids

Exclusion Criteria:

* Diagnosed neurological disease - eg Parkinson's disease, multiple sclerosis
* Cognitive impairment and dementia
* Bone fractures or joint replacement (in the past year)
* Pre-existing medical conditions from which the medical practitioner has advised not to exercise

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-11-19 (Actual); Study Completion 2023-11-19 (Actual)

PRIMARY OUTCOMES:
Laboratory induced falls | 12 month re-assessment
  Fall incidence after slips and trips in the laboratory (Okubo et al., 2019). A fall will be defined by the harness supported load when it exceeded 30% of the person's body weight (Yang et al., 2011).
Trips in daily life | Throughout a follow-up period (one year from randomisation)
  Number of trips in daily life will be recorded using a fridge calendar and reported weekly via SMS or email.
Slips in daily life | Throughout a follow-up period (one year from randomisation)
  Number of slips in daily life will be recorded using a fridge calendar and reported weekly via SMS or email.

SECONDARY OUTCOMES:
Falls in daily life | Throughout a follow-up period (one year from randomisation)
  Number of falls in daily life will be recorded using a fridge calendar and reported weekly via SMS or email.
Fall Risk | 12 month re-assessment
  A summary fall risk score will be calculated from the Physiological Profile Assessment short form which includes tests of vision, balance, proprioception, reaction time and strength (Lord et al., 2003).
Fear of falling | Week 3 (following the third training session)
  Fear of falling will be assessed using the Falls Efficacy Scale - International (Yardley et al., 2005), a 16 item scale scored out of 64 where higher scores indicate greater fear of falling
Fear of falling | Month 6 (middle of the follow-up period)
  Fear of falling will be assessed using the Falls Efficacy Scale - International (Yardley et al., 2005), a 16 item scale scored out of 64 where higher scores indicate greater fear of falling
Fear of falling | 12 month re-assessment
  Fear of falling will be assessed using the Falls Efficacy Scale - International (Yardley et al., 2005), a 16 item scale scored out of 64 where higher scores indicate greater fear of falling
Fall risk awareness and behaviours | Week 3 (following the third training session)
  Fall risk awareness and behaviours will be assessed using the 24-item Fall Behavioural Scale (Clemson et al., 2008). Mean scores range from 1.0 to 4.0 in which higher scores indicate safer behaviours
Fall risk awareness and behaviours | Month 6 (middle of the follow-up period)
  Fall risk awareness and behaviours will be assessed using the 24-item Fall Behavioural Scale (Clemson et al., 2008). Mean scores range from 1.0 to 4.0 in which higher scores indicate safer behaviours
Fall Behavioural Scale | 12 month re-assessment
  Fall risk awareness and behaviours will be assessed using the 24-item Fall Behavioural Scale (Clemson et al., 2008). Mean scores range from 1.0 to 4.0 in which higher scores indicate safer behaviours
Anxiety | 12 month re-assessment
  Anxiety will be assessed using the General Anxiety Disorder - 7-item scale (Spitzer, 2006), a 21 point scale where higher scores indicate greater anxiety
Physical activity levels | 12 month re-assessment
  Physical activity levels will be assessed using the Incidental and Planned Exercise Questionnaire (Delbaere et al., 2009). A total physical activity (hours per week) in the past 3 months will be estimated.
Volitional Stepping Reaction time | 12 month re-assessment
  Volitional stepping will be assessed using the Choice Stepping Reaction Time test standard version (Lord et al., 2001).
Stepping inhibition | 12 month re-assessment
  Stepping inhibition will be assessed using the Choice Stepping Reaction Time test moving arrow version.
Catch-inhibition accuracy | 12 month re-assessment
  Catch-inhibition accuracy will be assessed using the React Stick simple and complex modes (Richardson et al., 2017).
Executive function | 12 month re-assessment
  Executive function will be assessed using the Trail Making Test A and B (Tombaugh et al., 2004). Test scores B - A will be used as a measure of executive function.
Margin of stability | 12 month re-assessment
  Margin of stability (Hof et al., 2005) during the slip and trip trials will be assessed using the Vicon 3D motion analysis system with the full-body 27-marker model
Extrapolated centre of mass | 12 month re-assessment
  Extrapolated centre of mass (Hof et al., 2005) during the slip and trip trials will be assessed using the Vicon 3D motion analysis system with the full-body 27-marker model
Step length | 12 month re-assessment
  Step length during the slip and trip trials will be assessed using the Vicon 3D motion analysis system with the full-body 27-marker model
Range of trunk sway | 12 month re-assessment
  Range of trunk sway during the slip and trip trials will be assessed using the Vicon 3D motion analysis system with the full-body 27-marker model
Muscle activation onset latency (semitendinosus) | 12 month re-assessment
  Time (milliseconds) from a trip/slip onset to muscle activation onset will be recorded using surface electromyography on the semitendinosus. Muscle activation onset will be defined when the activation level exceeds 3 standard deviation above the baseline level.
Muscle activation onset latency (rectus femoris) | 12 month re-assessment
  Time (milliseconds) from a trip/slip onset to muscle activation onset will be recorded using surface electromyography on the rectus femoris. Muscle activation onset will be defined when the activation level exceeds 3 standard deviation above the baseline level.
Muscle activation amplitude (semitendinosus) | 12 month re-assessment
  Muscle activation amplitude will be recorded using surface electromyography on the semitendinosus. This will be assessed as percentage of the activation level during the trip and slip trials relative to the maximal voluntary contraction.
Muscle activation amplitude (rectus femoris) | 12 month re-assessment
  Muscle activation amplitude will be recorded using surface electromyography on the rectus femoris. This will be assessed as percentage of the activation level during the trip and slip trials relative to the maximal voluntary contraction.
Enjoyment of reactive balance training | Throughout training sessions taking place at week 1, 2 and 3, and month 3, 6 and 9
  Enjoyment of reactive balance training will be assessed using the 8-item Physical Activity Enjoyment Scale (PACES-8, Mullen et al., 2011). Scores range from 8 to 56 with higher scores indicate greater enjoyment.
Adverse events during reactive balance training | Throughout training sessions taking place at week 1, 2 and 3, and month 3, 6 and 9
  Adverse events such as muscle soreness, discomfort, pain or injury will be collected by staff during reactive balance training sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lord, PhD, Principal Investigator — Neuroscience Research Australia (NeuRA)
Locations (1):
- Neuroscience Research Australia, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data containing assessment results collected during the trial
Time Frame: Following publication of main study findings
Access Criteria: Request should be made to the principal investigator and UNSW Human Research Ethics Committee which will be reviewed on a case-by-case basis